CLINICAL TRIAL: NCT05830461
Title: Online Psychological Care Program to Reduce Psychological Distress in the Process of Diagnostic Evaluation and/or Screening of Mammary Glands in Women Who Attend a Breast Clinic.
Brief Title: Online Psychological Care Program for Women Who Attend a Breast Clinic.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Guadalajara (Other)
Collaborators: Instituto Mexicano del Seguro Social (Other Government); Tecnologico de Monterrey (Other); Universidad Internacional del Ecuador (Other); University of Twente (Other)
Responsible Party: Principal Investigator, Reyna Jazmin Martinez Arriaga, Principal Investigator, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CI-01022
Record Dates: First submitted 2023-03-21; First posted 2023-04-26 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer
Keywords: Cancer Screening Tests; Anxiety; Depression; Sense of coherence; Psychological Intervention; Internet-Based Intervention
MeSH Terms: conditions — Breast Neoplasms; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: The study has two arms, one is the experimental group that will receive the treatment through the online platform only, and the other is the comparison group that will receive the treatment delivered through printed visual material. The program consists of three stages that are aimed at: 1) Patients who undergo screening and obtain negative results for malignancy, 2) patients with suspicion and undergo a biopsy, 3) Patients with positive results for breast cancer.
Who Masked: Participant
Masking Description: The patients are not aware that there is an experimental group and a control group, the participants are not related and do not know each other.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group will receive the self-applied intervention through a digital platform. The intervention consists of three stages, depending on the situation of the patient: 1) Patients who undergo screening and obtain negative results for malignancy, 2) patients with suspicion and undergo a biopsy, 3) Patients with positive results for breast cancer.
  Interventions: Behavioral: Online psychological care program to reduce psychological distress in women who attend a breast clinic
- Control group (Active Comparator): The experimental group will receive the self-applied intervention through written visual material that will be given to them. The content of the material will be the same as the experimental group.
  Interventions: Behavioral: Psychological care program to reduce psychological distress in women who attend a breast clinic

INTERVENTIONS:
Behavioral: Online psychological care program to reduce psychological distress in women who attend a breast clinic — The intervention will be online and self-applied. It will consist of 3 stages, according to the patient's situation: 1) without suspicion of cancer (A1), 2) with suspicion of cancer (A2), and 3) with confirmed diagnosis of cancer (B).
  Stage 1 includes modules related to the prevention and timely detection of breast cancer. Stage A2 consists of emotional management in the face of suspicion of breast cancer. In stage B, medical information about breast cancer is provided, as well as psychological strategies to face the diagnosis.
  Psychological techniques based on the cognitive behavioral model, mindfulness, acceptance and commitment therapy, and health beliefs are included.
  Arms: Experimental group
Behavioral: Psychological care program to reduce psychological distress in women who attend a breast clinic — The intervention will be delivered through printed materials. It will consist of 3 stages, according to the patient's situation: 1) without suspicion of cancer (A1), 2) with suspicion of cancer (A2), and 3) with confirmed diagnosis of cancer (B).
  Stage 1 includes modules related to the prevention and timely detection of breast cancer. Stage A2 consists of emotional management in the face of suspicion of breast cancer. In stage B, medical information about breast cancer is provided, as well as psychological strategies to face the diagnosis.
  Psychological techniques based on the cognitive behavioral model, mindfulness, acceptance and commitment therapy, and health beliefs are included.
  Arms: Control group

SUMMARY:
The objective of this study is to evaluate the effectiveness of an online psychological care program to reduce anxiety, depression and negative psychological consequences and to increase a sense of coherence in the process of diagnostic evaluation and/or screening of mammary glands in women who attend a breast clinic.

There will be an experimental group and a control group. The experimental group will receive the psychological intervention through a virtual platform and the control group will be given visual material with the information. This platform will be designed based on the principles of user experience (UX).

DETAILED DESCRIPTION:
It has been shown that women who undergo diagnostic tests or screening of their mammary glands present symptoms associated with anxiety, concerns regarding a possible positive result for malignancy, as well as emotional distress. It is important to generate psychological programs aimed at reducing the psychological consequences of the diagnostic evaluation and/or screening of mammary glands because there are few approaches on the subject.

In Mexico there are breast clinics of the Mexican Social Security Institute, designed to perform screening tests and diagnostic evaluation of mammary glands, with the aim of identifying cases of breast cancer in early stages. However, few psychological interventions have been reported during the diagnostic process, so it is important to know the psychological affectations presented by women who undergo these tests. Given this, this intervention has the objective of evaluating the effectiveness of an online psychological care program to reduce psychological distress and increase the sense of coherence in the process of diagnostic evaluation of mammary glands in women who attend a breast clinic.

In the intervention there will be two groups: a) experimental group and b) control group.

The experimental group will receive online psychological care through the virtual platform and the patients in the control group will be given visual material with the information.

All participants will be invited to attend the breast clinic and undergo screening studies and/or diagnostic evaluation. For the assignment of the experimental and control group, it will be carried out through a randomization process through the Excel program.

ELIGIBILITY:
Inclusion Criteria:

* Patients of legal age who attend a health institution for screening studies and/or diagnostic evaluation of breast cancer.
* Patients who can use an electronic device (smart phone, computer, laptop, tablet) to access the virtual platform.
* Patients who give their informed consent to participate in the study.

Exclusion Criteria:

* Patients with suicidal ideation and/or attempt.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-19 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Change in the scores of the Hospital Anxiety and Depression Scale | 1 month, depends on when the participant finishes the modules.
  This is an instrument that comprises 14 items: seven to measure anxiety and seven to measure depression experienced in the previous week. The Hospital Anxiety and Depression Scale was validated in Mexican population with a reliability of 0.81 for anxiety and 0.82 for depression. Anxiety items evaluate whether the person has been worried or has experienced sensations of fear, while depression items evaluate anhedonia or pessimistic thoughts.
Change in the scores of the Psychological Consequences Questionnaire | 1 month, depends on when the participant finishes the modules.
  Evaluates the negative psychological consequences of breast cancer screening. It contemplates three dimensions: Emotional Affects, Physical Affects and Social Affects.

SECONDARY OUTCOMES:
Change in the scores of the Sense of coherence | 1 month, depends on when the participant finishes the modules.
  Evaluates coping with stressors in the illness-well-being continuum and possible solutions to the conflict. It contemplates three dimensions: understandability, manageability and significance. Reliability tests showed a Cronbach´s alpha of .80 overall scale in latin populations.

CONTACTS AND LOCATIONS:
Overall Officials: Reyna J Martínez Arriaga, PhD, Principal Investigator — University of Guadalajara; Alejandro Domínguez Rodríguez, PhD, Study Chair — University of Twente; Sergio O Meza Chavolla, MD, Study Chair — Instituto Mexicano del Seguro Social; Fabiola Macías Espinoza, PhD, Study Chair — University of Guadalajara; Joel O González Cantero, PhD, Study Chair — University of Guadalajara; Leivy P González Ramírez, PhD, Study Chair — Tecnologico de Monterrey; Paulina Herdoiza Arroyo, PhD, Study Chair — Universidad Internacional del Ecuador; Yineth A Muñoz Anacona, BD, Study Chair — University of Guadalajara
Locations (1):
- Instituto Mexicano del Seguro Social, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No
The participants will be recruited in a public health institution. Since it is a government institution, one of the rules regarding the information collected is that it cannot be shared with other people or institutions outside the institution.

REFERENCES:
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Cockburn J, De Luise T, Hurley S, Clover K. Development and validation of the PCQ: a questionnaire to measure the psychological consequences of screening mammography. Soc Sci Med. 1992 May;34(10):1129-34. doi: 10.1016/0277-9536(92)90286-y. PMID 1641674
- [Background] Antonovsky A. The structure and properties of the sense of coherence scale. Soc Sci Med. 1993 Mar;36(6):725-33. doi: 10.1016/0277-9536(93)90033-z. PMID 8480217
- [Background] Brandon CJ, Mullan PB. Patients' perception of care during image-guided breast biopsy in a rural community breast center: communication matters. J Cancer Educ. 2011 Mar;26(1):156-60. doi: 10.1007/s13187-010-0178-7. PMID 21188664
- [Background] Castaneda SF, Malcarne VL, Foster-Fishman PG, Davidson WS, Mumman MK, Riley N, Sadler GR. Health care access and breast cancer screening among Latinas along the California-Mexican border. J Immigr Minor Health. 2014 Aug;16(4):670-81. doi: 10.1007/s10903-013-9938-x. PMID 24150421
- [Background] Chujo M, Kigawa J, Okamura H. Psychological Factors and Characteristics of Recurrent Breast Cancer Patients with or without Psychosocial Group Therapy Intervention. Yonago Acta Med. 2011 Dec;54(4):65-74. Epub 2011 Dec 1. PMID 24031131
- [Background] Consedine NS, Magai C, Krivoshekova YS, Ryzewicz L, Neugut AI. Fear, anxiety, worry, and breast cancer screening behavior: a critical review. Cancer Epidemiol Biomarkers Prev. 2004 Apr;13(4):501-10. PMID 15066912
- [Background] Dominguez-Rodriguez A, Martinez-Luna SC, Hernandez Jimenez MJ, De La Rosa-Gomez A, Arenas-Landgrave P, Esquivel Santovena EE, Arzola-Sanchez C, Alvarez Silva J, Solis Nicolas AM, Colmenero Guadian AM, Ramirez-Martinez FR, Vargas ROC. A Self-Applied Multi-Component Psychological Online Intervention Based on UX, for the Prevention of Complicated Grief Disorder in the Mexican Population During the COVID-19 Outbreak: Protocol of a Randomized Clinical Trial. Front Psychol. 2021 Mar 29;12:644782. doi: 10.3389/fpsyg.2021.644782. eCollection 2021. PMID 33854466
- [Background] Fang SY, Wang YL, Lu WH, Lee KT, Kuo YL, Fetzer SJ. Long-term effectiveness of an E-based survivorship care plan for breast cancer survivors: A quasi-experimental study. Patient Educ Couns. 2020 Mar;103(3):549-555. doi: 10.1016/j.pec.2019.09.012. Epub 2019 Sep 12. PMID 31558323
- [Background] Galiano-Castillo N, Cantarero-Villanueva I, Fernandez-Lao C, Ariza-Garcia A, Diaz-Rodriguez L, Del-Moral-Avila R, Arroyo-Morales M. Telehealth system: A randomized controlled trial evaluating the impact of an internet-based exercise intervention on quality of life, pain, muscle strength, and fatigue in breast cancer survivors. Cancer. 2016 Oct 15;122(20):3166-3174. doi: 10.1002/cncr.30172. Epub 2016 Jun 22. PMID 27332968
- [Background] Hollis C, Morriss R, Martin J, Amani S, Cotton R, Denis M, Lewis S. Technological innovations in mental healthcare: harnessing the digital revolution. Br J Psychiatry. 2015 Apr;206(4):263-5. doi: 10.1192/bjp.bp.113.142612. PMID 25833865
- [Background] Holtdirk F, Mehnert A, Weiss M, Meyer B, Watzl C. Protocol for the Optimune trial: a randomized controlled trial evaluating a novel Internet intervention for breast cancer survivors. Trials. 2020 Jan 29;21(1):117. doi: 10.1186/s13063-019-3987-y. PMID 31996235
- [Background] Liao MN, Chen MF, Chen SC, Chen PL. Uncertainty and anxiety during the diagnostic period for women with suspected breast cancer. Cancer Nurs. 2008 Jul-Aug;31(4):274-83. doi: 10.1097/01.NCC.0000305744.64452.fe. PMID 18600114
- [Background] Montgomery M, McCrone SH. Psychological distress associated with the diagnostic phase for suspected breast cancer: systematic review. J Adv Nurs. 2010 Nov;66(11):2372-90. doi: 10.1111/j.1365-2648.2010.05439.x. PMID 21039773
- [Derived] Martinez-Arriaga RJ, Dominguez-Rodriguez A, Meza-Chavolla SO, Munoz-Anacona YA, Cisneros-Hernandez AA, Gonzalez-Cantero JO, Gonzalez-Ramirez LP, Herdoiza-Arroyo PE, Ruvalcaba-Romero NA, Macias-Espinoza F, Jimenez S. "Salud Mamaria", an internet-based psychoeducational program during the breast cancer diagnosis process: Protocol for a randomized controlled trial. Contemp Clin Trials Commun. 2024 Nov 26;43:101397. doi: 10.1016/j.conctc.2024.101397. eCollection 2025 Feb. PMID 39802661
- See also: Information about breast cancer screening — https://www.cancer.gov/espanol/tipos/seno/paciente/deteccion-seno-pdq

DOCUMENTS (1):
  • Informed Consent Form (2023-03-21): https://cdn.clinicaltrials.gov/large-docs/61/NCT05830461/ICF_000.pdf